CLINICAL TRIAL: NCT00156104
Title: A Multicenter, Randomized, Double-Blind, Fixed-Dose, 6-Week Trial of the Efficacy and Safety of Asenapine Compared With Placebo Using Haloperidol Positive Control in Subjects With an Acute Exacerbation of Schizophrenia
Brief Title: Efficacy and Safety of Asenapine With Placebo and Haloperidol (41023)(P05926)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05926; Hera; 41023
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Asenapine 5 mg BID
  Interventions: Drug: Asenapine
- 2 (Experimental): Asenapine 10 mg BID
  Interventions: Drug: Asenapine
- 3 (Active Comparator): Haloperidol 4m mg BID
  Interventions: Drug: Haloperidol
- 4 (Placebo Comparator): placebo
  Interventions: Other: Placebo arm

INTERVENTIONS:
Drug: Asenapine — 5 mg BID
  Arms: 1
Drug: Asenapine — 10 mg BID
  Arms: 2
Drug: Haloperidol — 4 mg BID
  Arms: 3
Other: Placebo arm
  Arms: 4

SUMMARY:
Schizophrenia is a brain disease. The primary features of schizophrenia are characterized by Positive symptoms (symptoms that should not be there, inability to think clearly, to distinguish reality from fantasy i.e., hearing voices) and Negative symptoms (a reduction or absence of normal behaviors or emotions, i.e., unable to manage emotions, make decisions and relate to others). Other symptoms include reduced ability to recall and learn new information, difficulty with problem solving, or maintaining productive employment. The symptoms of schizophrenia may be due to an imbalance in chemicals in the brain, primarily dopamine and serotonin, which enables brain cells to communicate with each other.

Asenapine is an investigational drug that may help to correct the inbalance in dopamine and serotonin. This is a 6-week trial to test the efficacy and safety of asenapine, compared with placebo, using an active comparator agent (haloperidol) in the treatment of patients with an acute exacerbation of schizophrenia. Patients who complete the 6-week trial will have the option of continuing in an additional one year extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Currently suffering from an acute exacerbation of schizophrenia. Caregiver required.

Exclusion Criteria:

* Have an uncontrolled, unstable medical condition. Have any other pyschiatric disorder other than schizophrenia as a primary diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2005-07-01 (Actual); Primary Completion 2006-08-18 (Actual); Study Completion 2006-09-16 (Actual)

PRIMARY OUTCOMES:
Improvement in schizophrenia (change in total PANSS score) from baseline to endpoint (LOCF/MMRM) | Primary outcome measured weekly for 6 weeks

SECONDARY OUTCOMES:
Other dimensions of schizophrenia (positive, negative, disorganized thought, hostility/excitement, anxiety/depression, and general psychopathology) CGI-S; CGI-I | At weekly intervals throughout the 6-week trial.
Neurocognition and cognitive functioning | Baseline and Endpoint ( Day 42)
CDSS | Days 21 and 42(Endpoint).
Suicidal thinking ( ISST modified) | Days 14 and 42 (Endpoint)
Quality of life and patient functionality (QLS; Q-LES-Q ;PETIT0; Physical exam; Pregnancy test | Baseline and Day 42(Endpoint)
Readiness to discharge | At weekly intervals during the 6-week trial
EPS ( AIMS; BARS; SARS) | At weekly intervals during the 6-week triaL
Labs; Vital Signs; Weight and girth; ECG | Days 14; 28 and 42 (Endpoint)
Safety and Tolerability

REFERENCES:
- [Result] Kane JM, Cohen M, Zhao J, Alphs L, Panagides J. Efficacy and safety of asenapine in a placebo- and haloperidol-controlled trial in patients with acute exacerbation of schizophrenia. J Clin Psychopharmacol. 2010 Apr;30(2):106-15. doi: 10.1097/JCP.0b013e3181d35d6b. PMID 20520283
- [Derived] Castle DJ, Slott Jensen JK. Management of depressive symptoms in schizophrenia. Clin Schizophr Relat Psychoses. 2015 Apr;9(1):13-20. PMID 25367164